CLINICAL TRIAL: NCT05772702
Title: Closed-Loop Transcranial Alternating Current Stimulation for the Treatment of Depression (CLACS): Single-Site Open-Label Pilot Study
Brief Title: Closed-Loop Transcranial Alternating Current Stimulation for the Treatment of Depression
Acronym: CLACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Electromedical Products International, Inc. (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-3094
Record Dates: First submitted 2023-02-24; First posted 2023-03-16 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Depression; Major Depressive Disorder; tACS
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Closed-loop tACS (Experimental): Closed-loop individual alpha tACS daily for five consecutive days.
  Interventions: Device: Closed-loop tACS

INTERVENTIONS:
Device: Closed-loop tACS — Individual alpha tACS

SUMMARY:
The purpose of this research study is to study closed-loop transcranial alternating current stimulation (tACS) to determine its effects on symptoms of depression in people with major depressive disorder.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to investigate the preliminary efficacy of closed-loop tACS for the treatment of major depressive disorder (MDD) in an open-label pilot study. We will recruit up to 35 participants with unipolar, non-psychotic MDD. Participation will include seven visits, two of them remotely (with an in-person option as needed), and one electronic survey.

Potential participants fill-in an electronic pre-screening form. If potentially eligible, a remote screening visit is performed. If eligible, participants attend five consecutive, daily stimulation sessions. Clinical assessments will be performed at baseline (Day 1 of stimulation, D1), Day five of stimulation (D5), and at their follow-up visit (14 days after the completion of stimulation, FU2) using the Hamilton Depression Rating Scale (HDRS-17).

For a subset of patients, electroencephalography (EEG) is collected at D1 prior to stimulation and after stimulation and again at FU2.

For a subset of patients, self-scoring surveys will be sent bi-weekly until 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* Diagnostic and Statistical Manual, 5th Edition (DSM-5) diagnosis of MDD; unipolar, non-psychotic
* Hamilton Rating Depression Rating Scale (HRDS-17) score >8
* Low suicide risk as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) triage form (no intent or plan)
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)

Exclusion Criteria:

* DSM-5 diagnosis of severe alcohol use disorder (AUD) within the last 12 months.
* DSM-5 diagnosis of moderate to severe substance use disorder (excluding tobacco) within the last 12 months.
* Lifetime history of bipolar disorder, psychotic disorder, schizophrenia, autism
* Current use of benzodiazepines > 20mg diazepam/d equivalent
* Antidepressant dose change within the last 2 weeks
* Initiated new antidepressant within the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Rubinow, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander ML, Alagapan S, Lugo CE, Mellin JM, Lustenberger C, Rubinow DR, Frohlich F. Double-blind, randomized pilot clinical trial targeting alpha oscillations with transcranial alternating current stimulation (tACS) for the treatment of major depressive disorder (MDD). Transl Psychiatry. 2019 Mar 5;9(1):106. doi: 10.1038/s41398-019-0439-0. PMID 30837453
- See also: Link to more information and study recruitment for interested potential participants. — https://researchforme.unc.edu/index.php/en/study-details?rcid=4419

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed-loop tACS
Started | 26 (One participant experienced nausea and vomiting during the first treatment session. These transient symptoms were deemed to be mild and considered unlikely to be related to stimulation by the study clinician since the participant did not disclose an ongoing COVID-19 infection, which included headache, dizziness, and nausea before stimulation onset. Study participation was ended for this participant.)
Completed | 25
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (15.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20
  Male | 4
  Gender nonconforming | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 4
  Unknown or Not Reported | 0
Baseline HDRS-17 Score [Mean (Standard Deviation); unit: units on a scale] — Baseline HDRS-17 (Hamilton Depression Rating Scale, 17-item) score on Day 1 (D1) of treatment week prior to receiving treatment; minimum value is 0, maximum value is 52. Higher scores indicate worse outcome.
  units on a scale | 17.18 (4.19)
Baseline QIDS Score [Mean (Standard Deviation); unit: units on a scale] — Baseline QIDS (Quick Inventory of Depressive Symptomatology) score on Day 1 (D1) of treatment week prior to receiving treatment; minimum value is 0, maximum value is 27. Higher scores indicate worse outcome.
  units on a scale | 14.72 (2.67)
Baseline Q-LES-Q-SF Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Q-LES-Q-SF (Quality of Life Enjoyment and Satisfaction Questionnaire, Short Form) on day 1 (D1); minimum value is 14, maximum value is 70. Higher scores indicate better outcome.
  units on a scale | 37.44 (5.12)
Baseline ASRM Score [Mean (Standard Deviation); unit: units on a scale] — Baseline ASRM (Altman Self-Rating Mania Scale) on day 1 (D1); minimum value is 0, maximum value is 20. Higher scores indicate worse outcome.
  units on a scale | 1.16 (1.28)
Baseline SHAPS Score [Mean (Standard Deviation); unit: units on a scale] — Baseline SHAPS (Snaith-Hamilton Pleasure Scale) score on day 1 (D1); minimum value is 0, maximum value is 14. Higher scores indicate worse outcome.
  units on a scale | 5.52 (3.27)
Baseline DASS-42 Score [Mean (Standard Deviation); unit: units on a scale] — Baseline DASS-42 (Depression, Anxiety, and Stress Scale, 42-item) on day 1 (D1); minimum value is 0, maximum value is 126 with three subscales (0 to 42). Higher scores indicate worse outcome.
  units on a scale
    Overall Score | 45.96 (14.42)
    Depression Subscale | 23.12 (6.31)
    Anxiety Subscale | 6.48 (4.09)
    Stress Subscale | 16.36 (9.34)
Baseline STAI Score [Mean (Standard Deviation); unit: units on a scale] — Baseline STAI (State-Trait Anxiety Inventory (state score)) on day 1 (D1); minimum value is 20, maximum value is 80. Higher scores indicate worse outcome.
  units on a scale | 47.88 (10.78)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale 17-item (HDRS-17)
Description: Change in HDRS-17 from Day 1 (D1) to Day 19 (i.e., two week follow-up; FU2); HDRS-17 minimum value is 0, maximum value is 52. Higher scores indicate worse outcome. Negative scores indicate improved outcomes.
Time Frame: Day 1 to Day 19 (i.e. 19 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
units on a scale | -12.04 (4.83)
Statistical Analysis 1: Comparison: Closed-loop tACS; HDRS-17 change score were submitted to a t-test to estimate the group difference from 0 (i.e., no change in depression symptoms from D1 to FU2). Null hypothesis: D1 == FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, t-test, 2 sided

2. Secondary Outcome: Change in Hamilton Depression Rating Scale 17-item (HDRS-17)
Description: Change in HDRS-17 from Day 1 (D1) to Day 5 (D5); HDRS-17minimum value is 0, maximum value is 52. Higher scores indicate worse outcome. Negative scores indicate improved outcomes.
Time Frame: Day 1 to Day 5 (i.e., 5 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale | -8.36 (4.41)
Statistical Analysis 1: Comparison: Closed-loop tACS; HDRS-17 change score were submitted to a t-test to estimate the group difference from 0 (i.e., no change in depression symptoms from D1 to D5). Note: D5 HDRS-17 were determined prior to receiving the final treatment on D5. Null hypothesis: D1 == D5; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, t-test, 2 sided

3. Secondary Outcome: Response/Remission of Depression
Description: Number of response/remission rates at Day 5 (D5) and Day 19 (i.e., two week follow-up; FU2). Response defined as >=50% reduction in HDRS-17 from D1. Remission defined as HDRS-17 score <=7.
Time Frame: Day 5 and Day 19
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
Participants
  Response at D5: Met criteria | 12
  Response at D5: Did not meet criteria | 13
  Response at FU2: Met criteria | 21
  Response at FU2: Did not meet criteria | 4
  Remission at D5: Met criteria | 10
  Remission at D5: Did not meet criteria | 15
  Remission at FU2: Met criteria | 21
  Remission at FU2: Did not meet criteria | 4

4. Secondary Outcome: Change in Quick Inventory of Depressive Symptomatology (QIDS)
Description: Change in QIDS at Day 5 (D5), Day 12 (i.e., one-week follow-up; FU1), and Day 19 (i.e., two-week follow-up; FU2); QIDS minimum value is 0, maximum value is 27. Higher scores indicate worse outcome. Negative scores indicate improved outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  D5-D1 | -3.88 (3.23)
  FU1-D1 | -5.96 (3.51)
  FU2-D1 | -7.48 (3.90)
Statistical Analysis 1: Comparison: Closed-loop tACS; QIDS change score were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 QIDS surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; Mauchly's test of sphericity determined the sphericity assumption was violated, so Greenhouse-Geisser corrections were applied

5. Secondary Outcome: Change in Altman Self-Rating Mania Scale (ASRM)
Description: Change in ASRM at Day 5 (D5), Day 12 (i.e., one week follow-up; FU1), and Day 19 (i.e., two week follow-up; FU2); ASRM minimum value is 0, maximum value is 20. Higher scores indicate worse outcome. Negative scores indicate improved outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  D5-D1 | 0.88 (1.81)
  FU1-D1 | 1.92 (1.93)
  FU2-D1 | 1.92 (1.89)
Statistical Analysis 1: Comparison: Closed-loop tACS; ASRM scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 ASRM surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA

6. Secondary Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS)
Description: Change in SHAPS from Day 1 (D1) to Day 5 (D5), Day 12 (i.e., one week follow-up; FU1), and Day 19 (i.e., two week follow-up; FU2); SHAPS minimum value is 0, maximum value is 14. Higher scores indicate worse outcome. Negative scores indicate improved outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  D5-D1 | -2.60 (2.61)
  FU1-D1 | -3.48 (3.40)
  FU2-D1 | -3.76 (3.44)
Statistical Analysis 1: Comparison: Closed-loop tACS; SHAPS scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 SHAPS surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; [statistical method as in outcome 4, analysis 1]

7. Secondary Outcome: Change in Depression Anxiety and Stress Scale (DASS-42)
Description: Change in DASS-42 from Day 1 (D1) to Day 5 (D5), Day 12 (i.e., one week follow-up; FU1), and Day 19 (i.e., two week follow-up; FU2); DASS-42 minimum value is 0, maximum value is 126 with three subscales (0 to 42). Higher scores indicate worse outcome. Negative scores indicate improved outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  Overall: D5-D1 | -12.52 (14.39)
  Overall: FU1-D1 | -21.44 (16.63)
  Overall: FU2-D1 | -24.08 (18.92)
  Depression Subscale: D5-D1 | -6.52 (8.15)
  Depression Subscale: FU1-D1 | -11.00 (7.53)
  Depression Subscale: FU2-D1 | -12.20 (8.90)
  Anxiety Subscale: D5-D1 | -1.88 (2.57)
  Anxiety Subscale: FU1-D1 | -2.84 (4.04)
  Anxiety Subscale: FU2-D1 | -3.64 (4.51)
  Stress Subscale: D5-D1 | -4.12 (6.73)
  Stress Subscale: FU1-D1 | -7.60 (8.99)
  Stress Subscale: FU2-D1 | -8.24 (9.47)
Statistical Analysis 1: Comparison: Closed-loop tACS; DASS-42 OVERALL scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 DASS-42 surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Closed-loop tACS; DASS-42 DEPRESSION SUBSCORES were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 DASS-42 surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; This subscale did not require sphericity corrections
Statistical Analysis 3: Comparison: Closed-loop tACS; DASS-42 ANXIETY SUBSCORES were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 DASS-42 surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Closed-loop tACS; DASS-42 STRESS SUBSCORES were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 DASS-42 surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Change in State-Train Anxiety Inventory (STAI)
Description: Change in STAI from Day 1 (D1) to Day 5 (D5), Day 12 (one week follow-up; FU1), and Day 19 (two week follow-up; FU2); STAI minimum value is 20, maximum value is 80. Higher scores indicate worse outcome. Negative scores indicate improved outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  D5-D1 | -3.08 (10.03)
  FU1-D1 | -5.16 (10.35)
  FU2-D1 | -6.16 (12.29)
Statistical Analysis 1: Comparison: Closed-loop tACS; STAI scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 STAI surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p = 0.021, ANOVA; [statistical method as in outcome 4, analysis 1]

9. Secondary Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire, Short Form (Q-LES-Q-SF)
Description: Change in Q-LES-Q-SF from Day 1 (D1) to Day 5 (D5), Day 12 (i.e., one week follow-up; FU1), and Day 19 (i.e., two week follow-up; FU2); Q-LES-Q-SF minimum value is 14, maximum value is 70. Higher scores indicate better outcome. Negative scores indicate worse outcome.
Time Frame: Day 1 (D1) to Day 5 (D5); D1 to Day 12 (FU1); and D1 to Day 19 (FU2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
score on a scale
  D5-D1 | 6.86 (12.58)
  FU1-D1 | 15.36 (11.34)
  FU2-D1 | 16.57 (13.56)
Statistical Analysis 1: Comparison: Closed-loop tACS; QIDS scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 QIDS surveys were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU1 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA

10. Secondary Outcome: Change in Clinical Global Impression Scale (CGI)
Description: Change in CGI from Day 1 (D1) to Day 5 (D5) and Day 19 (i.e., two week follow-up; FU2); CGI scale contains two scoring components, 1) Severity of Illness (0-7) and 2) Global Improvement (0-7). Higher scores in component 1 indicate worse symptoms while higher numbers in component 2 indicate worse clinical outcomes.
Time Frame: Severity: {Day 1 (D1), Day 5 (D5) and Day 19 (FU2)}; Global Improvement: {Day 5 (D5) and Day 19 (FU2)}
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Closed-loop tACS
Number analyzed (Participants) | 25
units on a scale
  Global Improvement at D5 | 2.56 (1.16)
  Global Improvement at FU2 | 1.68 (0.75)
  Severity at D1 | 4.04 (0.79)
  Severity at D5 | 2.36 (1.19)
  Severity at FU2 | 1.76 (0.93)
Statistical Analysis 1: Comparison: Closed-loop tACS; CGI severity scores were submitted to a repeated measures ANOVA to measure change from baseline over time. Note: D5 CGI assessments were completed prior to receiving the final treatment on D5. Null hypothesis: D1 = D5 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p < 0.0005, ANOVA
Statistical Analysis 2: Comparison: Closed-loop tACS; CGI improvement scores were submitted to a paired t-test to measure difference between the improvement assessment on D5 and the assessment at FU2. Note: D5 CGI assessments were completed prior to receiving the final treatment on D5. Null hypothesis: D5 = FU2; Test type: Other — This was a single-arm, open-label trial. Reported statistics reflect changes from baseline levels; p = 0.006, t-test, 2 sided

11. Other Pre Specified Outcome: Change in Alpha Oscillation Power
Description: Change in EEG alpha oscillation power at D1 pre-stimulation, D1 post-stimulation, and FU2.
Time Frame: 19 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Quick Inventory of Depressive Symptomatology (QIDS) Over 12 Weeks
Description: Change in QIDS at four week follow-up (FU3), six week follow-up (FU4), eight week follow-up (FU5), ten week follow-up (FU6), and twelve week follow-up (FU7); minimum value is 0, maximum value is 27. Higher scores indicate worse outcome.
Time Frame: 89 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Altman Self-Rating Mania Scale (ASRM) Over 12 Weeks
Description: Change in ASRM at FU3, FU4, FU5, FU6, and FU7; minimum value is 0, maximum value is 20. Higher scores indicate worse outcome.
Time Frame: 89 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS) Over 12 Weeks
Description: Change in SHAPS at FU3, FU4, FU5, FU6, and FU7; minimum value is 0, maximum value is 14. Higher scores indicate worse outcome.
Time Frame: 89 days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in Depression Anxiety and Stress Scale (DASS-42) Over 12 Weeks
Description: Change in DASS-42 at FU3, FU4, FU5, FU6, and FU7; minimum value is 0, maximum value is 126 with three subscales (0 to 42). Higher scores indicate worse outcome.
Time Frame: 89 days
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in State-Train Anxiety Inventory (STAI) Over 12 Weeks
Description: Change in STAI at FU3, FU4, FU5, FU6, and FU7; minimum value is 20, maximum value is 80. Higher scores indicate worse outcome.
Time Frame: 89 days
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire, Short Form (Q-LES-Q-SF)
Description: Change in Q-LES-Q-SF at FU3, FU4, FU5, FU6, and FU7; minimum value is 14, maximum value is 70. Higher scores indicate better outcome.
Time Frame: 89 days
Reporting Status: Not Posted

18. Other Pre Specified Outcome: HDRS-17 Change
Description: Change in HDRS-17 between six week follow up (FU4) and D1
Time Frame: 47 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected across the full study participation (89 days). A structured adverse event was administered on D5 for all participants and for any AE spontaneously reported by a participant.
Arm/Group | Closed-loop tACS
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 21/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-loop tACS (N=26)
Nausea (Gastrointestinal disorders) | 2 (2) — Nausea, time-limited to the stimulation session
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting, time-limited to the stimulation session, determined by study physician to likely be related to participant's undisclosed COVID-19 infection.
Diarrhea (Gastrointestinal disorders) | 3 (3) — Diarrhea reported during the treatment week
Headache (Nervous system disorders) | 13 (13) — Headache, time-limited to the stimulation session
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) — Skin irritation at electrode sites, time-limited to the stimulation session
Scalp/neck pain (General disorders) | 2 (2) — Scalp/neck pain, time-limited to the stimulation session
Dizziness (Nervous system disorders) | 2 (2) — Dizziness, time-limited to the stimulation session
Fatigue (General disorders) | 13 (13) — Fatigue, increased tiredness time-limited to the stimulation session
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle cramps, time-limited to the stimulation session

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT05772702/Prot_SAP_000.pdf